CLINICAL TRIAL: NCT02941146
Title: DualSculpting the Abdomen Using CoolSculpting
Acronym: DSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA16-004
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Results first posted 2020-12-21 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2016-10

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Zeltiq Dual Sculpting Treatment Group (Experimental): All subjects treated with CoolSculpting System using the CoolAdvantage and CoolAdvantage Plus applicators simultaneously on the abdomen.
  Interventions: Device: The ZELTIQ System

INTERVENTIONS:
Device: The ZELTIQ System — The CoolSculpting System will be used to perform the treatments with the CoolAdvantage family of applicators.

SUMMARY:
Evaluate the safety and efficacy of abdominal DualSculpting with CoolAdvantage applicators.

DETAILED DESCRIPTION:
The study will evaluate the safety and efficacy of non-invasive fat reduction in the abdomen using two applicators.

ELIGIBILITY:
Inclusion Criteria

1. Male or female subjects >22 years of age and < 65 years of age.
2. Subject who has been assessed to be eligible to receive multiple DualSculpting treatments on the abdomen using the CoolAdvantage and/or CoolAdvantage Plus applicator.
3. No weight change exceeding 5% of body weight in the preceding month.
4. Subject agrees to maintain his/her weight (i.e., within 5%) by not making any major changes in their diet or exercise routine during the course of the study.
5. Subject has read and signed the study written informed consent form.

Exclusion Criteria

1. Subject has had a surgical procedure(s) in the area of intended treatmentSubject has had a surgical procedure(s) in the area of intended treatment.
2. Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
3. Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 12 months.
4. Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
5. Subject has a known history of cryoglobulinemia, cold urticaria, cold agglutinin disease or paroxysmal cold hemoglobinuria.
6. Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
7. Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
8. Subject is taking or has taken diet pills or supplements within the past month.
9. Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
10. Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system or any other metal containing implant.
11. Subject is pregnant or intending to become pregnant during the study period
12. Subject is lactating or has been lactating in the past 6 months.
13. Subject has a history of hernia in the areas to be treated.
14. Subject is unable or unwilling to comply with the study requirements.
15. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
16. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Main Line Center for Laser Surgery, Ardmore, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol defined inclusion and exclusion conditions determined study entry. All subjects were included in the single arm study.
Groups:
- CoolSculpting of the Abdomen: Non-invasive fat reduction of the abdomen will be performed using the Zeltiq CoolSculpting System.
Period: Overall Study
Arm/Group | CoolSculpting of the Abdomen
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Candidates who sought reduction of fat in the abdomen and who the investigator has assessed to be eligible for multiple DualSculpting treatments in the abdomen were eligible to participate.
Groups:
- CoolSculpting of the Abdomen With Dual Applicators: Non-invasive fat reduction of the abdomen was performed using the Zeltiq CoolSculpting System using dual applicators.
Arm/Group | CoolSculpting of the Abdomen With Dual Applicators
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 0
  Asian | 0
  Hispanic | 0
  Caucasian | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 29.5 [25.5 to 36.7]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Correctly Identified Photos by Blinded Reviewers
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images. Reviewers will be practicing dermatologists or plastic surgeons. All reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which images will be presented will be randomized; for each subject placement of the baseline, pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. The primary efficacy endpoint of the study was the correct identification of baseline (pre-treatment) vs. 12 weeks post-final treatment images by two out of three blinded, independent reviewers. Success was defined as at least 70% correct identification of the baseline (pre-treatment) photographs.
Time Frame: Baseline to 12 weeks post-treatment
Population: Fourteen of 15 treated subjects were included in the per-protocol analysis. One subject was excluded from analysis due to a protocol-defined weight maintenance requirement. Pre-treatment and post-treatment photos were evaluated by 3 independent physician reviewers.
Measure: Count of Units; unit: photos
Units Other Than Participants: photos
Arm/Group | CoolSculpting of the Abdomen With Dual Applicators
Number analyzed (Participants) | 14
Number analyzed (photos) | 42
photos | 28
Statistical Analysis 1: Comparison: CoolSculpting of the Abdomen With Dual Applicators; Test type: Other; sucess proportion = 64.3, 95% CI 2-sided [35.1 to 87.2]

2. Primary Outcome: Safety of the Zeltiq Device
Description: The incidence of unanticipated adverse device effects will be measured. It is expected there will be zero UADEs.
Time Frame: 12 week post-treatment
Population: The "as-treated" population included all subjects who were treated with CoolSculpting.
Measure: Number; unit: device-or procedure-related AEs
Arm/Group | CoolSculpting of the Abdomen With Dual Applicators
Number analyzed (Participants) | 15
device-or procedure-related AEs | 0

3. Secondary Outcome: Subject Satisfaction
Description: Subject satisfaction with the Zeltiq procedure as determined by positive responses in a subject satisfaction questionnaire administered at the 12 weeks post-treatment visit. This questionnaire will be composed of 5-point Likert scale questions, as well as free-text responses, with lower numbers (e.g. 1 or 2) indicating positive responses and higher numbers indicating less positive responses.
Time Frame: 12 weeks post-treatment
Population: The per-protocol population consisted of 14 subjects. One subject was excluded for weight gain >5%, a protocol defined limit for weight maintenance and was excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CoolSculpting of the Abdomen With Dual Applicators
Number analyzed (Participants) | 14
Participants
  Procedure comfortable/very comfortable | 7
  Feel appearance improved | 8
  Satisfied or very satisfied with procedure | 9
  Would recommend to a friend | 7

ADVERSE EVENTS:
Time Frame: Adverse event data was solicited continuously throughout the study. The final follow-up visit occurred 12 weeks post-treatment.
Description: Adverse events (AE) will be assessed continuously throughout the study. An adverse event is defined as any untoward medical occurrence in a subject, regardless of whether the event is related to the device. Common minor health complaints related to the upper respiratory tract (e.g. rhinitis, influenza, common cold) will not be documented as adverse events.
Arm/Group | CoolSculpting of the Abdomen With Dual Applicators
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT02941146/Prot_SAP_000.pdf